CLINICAL TRIAL: NCT03296085
Title: A Simple Technique for Quantitative Evaluation of an Important Clinical Sign
Brief Title: Bedside Evaluation of Edema
Acronym: EDEMA
Status: Terminated | Type: Observational
Why Stopped: Principle investigator changed academic affiliation, then later retired. Study terminated after intra-observer validation, but inter-observer validation not completed.
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Richard Schreiber, MD FACP, Chief Medical Informatics Officer, Geisinger Clinic
Other Study IDs: 2017-0434
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Edema
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Exam for quantity of edema — There is no intervention

SUMMARY:
Edema, commonly called swelling, is a common medical condition, with many causes. Clinicians generally find edema by pressing against a patient's skin, usually on the feet or shins, and observing how much dimpling there is in the skin. Most clinicians estimate the amount on a scale of mild to severe, or perhaps state the amount as 1 to 4. There is little agreement between observers, and it is hard to judge different clinicians' use of these scales. The first part of this experiment will demonstrate this inconsistency. After clinicians are shown a new technique for measuring edema, the second part of the study will show more accurate and consistent measurements. This will help clinicians to measure edema better, and to communicate their findings to other clinicians more effectively.

DETAILED DESCRIPTION:
The research team will recruit as many clinicians who are conveniently available for the study. Clinicians will include attending physicians from any specialty, residents, medical students, physician assistants, physician assistant students, nurses, certified nurse practitioners, and certified nurse practitioner students.

Once patients and clinicians have been recruited, the research team will maintain a list of the patients and a grid of which clinicians are to examine which patients. Each clinician will be given a data collection sheet, listing the patients' room numbers, and a grid for recording results for each of the patient's affected limb(s). The first data collection sheet (before instruction on the quantitative method) will just show a blank free text field so that clinicians can record their results as they normally do.

After instruction in the novel quantitative technique, the clinicians will receive another data collection sheet now indicating the intent to have the clinicians record their findings in millimeters.

The expectation is that a minimum of 6 examiners will determine the extent of edema on at least 38 limbs. If possible, the research will continue until approximately 100 limbs have been examined by a total of at least 10 to 20 clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Currently admitted patients
* Patient who can understand the purpose of the study and sign a consent form
* Patient has a measurable amount of edema
* Patient will likely be available during the time the clinicians can examine the patient

Exclusion Criteria:

* Unable or unwilling to sign the consent form
* No measurable edema
* Currently in isolation for infection control purposes
* Patients in the Behavioral Health section of the hospital
* Maternity patients (due to availability of infant rooming-in)
* Prisoners
* Age below 18 years
* Patients with bilateral lower extremity amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with edema
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Inter-observer correlation of edema measurement before instruction in novel technique | one day
  Observe the variation in edema documentation based on standard examination technique
Inter-observer correlation of edema measurement after instruction in novel technique | one day
  Observe the variation in edema documentation based on the novel examination technique

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schreiber, MD, Principal Investigator — Geisinger Holy Spirit
Locations (1):
- Geisinger Holy Spirit, Camp Hill, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No